CLINICAL TRIAL: NCT01755481
Title: Feeding Infant Formula With Added Probiotics and Whey Protein Concentrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arla Foods (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 327727-2
Record Dates: First submitted 2012-12-12; First posted 2012-12-24 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Focus on Healthy Infants
MeSH Terms: interventions — Probiotics; Whey

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics F19 (Experimental): F19 in an infant formula
  Interventions: Other: Probiotic
- Whey protein concentrate (Experimental): Whey protein concentrate in an infant formula
  Interventions: Other: Whey protein concentrate

INTERVENTIONS:
Other: Probiotic
  Arms: Probiotics F19
Other: Whey protein concentrate
  Arms: Whey protein concentrate

SUMMARY:
To evaluate the effects of feeding an infant formula containing L. paracasei ssp. paracasei strain F19 or Whey Protein Concentrate.

ELIGIBILITY:
Inclusion criteria (formula-fed group):

healthy infants of mothers who could not or voluntarily resigned completely from breast-feeding at infant age 14 plus/minus 3 days

Inclusion criteria (breast-fed group):

healthy infants exclusively breast-fed from birth and mothers intending to breastfeed >80% until at least 5th month of age (meaning through the 4th month of age).

Inclusion criteria (all infants):

delivered between 37 and 42 weeks of gestation birth weight >2500 g and <4000 g parent or the subject's legal representative speak and understand Chinese

Exclusion criteria (formula-fed group):

fully or partially breast-fed infants infants breast-fed >20%

Exclusion criteria (breast-fed group):

infants fed >20% infant formula

Exclusion criteria (all infants):

malformations, handicaps or congenital diseases that could affect normal feeding or growth treatment with antibiotics

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2012-12; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Infections episodes (gastrointestinal and upper and lower respiratory infections) | 4 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Peng, M.D., Ph.D., Principal Investigator — Children's Hospital, Fudan University, Shanghai, China
Locations (1):
- Department of Child Health Care, Children's Hospital, Fudan University, Shanghai, China